CLINICAL TRIAL: NCT06777810
Title: Genetic Identification and Quantitative Analysis of Pathogenic Bacteria of Diabetic Foot Ulcer Infection
Brief Title: Identification of Pathogenic Bacteria of Diabetes Foot Ulcer
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Wang Weiqing, Professor, Ruijin Hospital
Other Study IDs: CCEMD-20241002
Record Dates: First submitted 2024-12-10; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-11

CONDITIONS: Diabetic Foot Disease; Diabetic Foot Ulcer; Diabetes
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: The infected wound of the patient's foot ulcer was collected — The infected wound of the patient's foot ulcer was collected

SUMMARY:
The objective of this study is to design and develop a gene chip for detecting pathogenic bacteria in diabetic foot infection wounds. This innovative gene chip technology enables rapid and accurate identification of pathogens at the site of infection by detecting the 16SrDNA sequence of pathogenic bacteria.

Diabetic foot infection is a common serious complication in diabetic patients, often accompanied by complex pathogenic bacteria population, and due to the variety of infection types, traditional pathogen detection methods are time-consuming and low accuracy, patients may miss the best treatment opportunity. Now commonly used genetic identification of pathogenic bacteria often find a variety of bacteria, resulting in the actual pathogenic bacteria difficult to judge.

DETAILED DESCRIPTION:
Based on the principle of 16SrDNA detection, this study developed an efficient and convenient gene chip, which can accurately identify and quantitatively analyze different types of pathogenic bacteria at the molecular level. Through this technology, it can significantly improve the diagnostic efficiency and accuracy of diabetic foot infection, provide patients with more timely treatment, reduce the risk of complications caused by infection, and improve the quality of life of patients.

Objective:

1. Development of efficient gene chip: Design a gene chip that can rapidly detect pathogenic bacteria in diabetic foot infection wounds. By detecting the 16SrDNA sequence, the chip can identify a variety of pathogenic bacteria and provide accurate data support for clinical diagnosis
2. Evaluate the difference in detection time between gene-chip detection technology and traditional schemes: traditional bacterial culture and identification methods usually take several days, but this study aims to shorten the detection time (i.e. the time from taking wound samples to getting pathogenic bacteria detection results) to several hours through gene-chip technology, so as to improve the diagnostic efficiency and obtain pathogenic bacteria information in time
3. Compare the sensitivity and specificity of gene chip and traditional methods (such as bacterial culture) in detecting pathogenic bacteria, and then obtain the changes in the diagnostic accuracy of gene chip technology: The Sensitivity, Specificity, positive predictive value (PPV), negative predictive value (NPV) and other key diagnostic indicators of the pathogen were tested for specificity of diabetic foot infection, and the diagnostic accuracy of specificity was verified by comparing with traditional bacterial specificity Methods:This study is a scientific research project carried out in the laboratory. Through consulting the common bacterial strains cultured by diabetic foot infection in our hospital, the probe is made by adding anaerobic bacterial strains according to the literature. Informed consent was signed, about 60 subjects were recruited according to inclusion and exclusion criteria, and more than three specimens were collected for each subject. One was used to analyze pathogenic bacteria by conventional bacterial culture method; One pathogen was sequenced using conventional 16SrDNA; A gene chip analysis, using quantitative chip technology, to determine the content of each bacteria, with the highest content of bacteria reference as a pathogen. The sequencing result of bacterial content detected by bacterial 16SrDNA chip, the highest content, should be consistent with the conventional bacterial culture results.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Gender: males and females
3. Patients diagnosed with diabetic foot infection with an infected wound
4. It can provide sufficient infected wound samples (≥5mm³ infected wound tissue samples or ≥100μL infected wound secretions) and can be used for detection and analysis of gene chips
5. No history of antibiotic therapy prior to sampling (within 4 weeks) or known failure to respond to antibiotic therapy (failure to respond to ≥2 antibiotics)
6. Fully understand the nature, significance, possible benefits, possible inconveniences or potential risks of this research; Understand the study procedure, participate voluntarily and be willing to complete the entire study process, and sign the informed consent

Exclusion Criteria:

1. Patients with undiagnosed diabetic foot infection
2. Patients who had received antibiotics within 4 weeks prior to sampling
3. Complicated with serious systemic disease (e.g., malignant tumor, severe cardiopulmonary insufficiency, etc.)
4. Pregnant or lactating women
5. Cognitive impairment or inability to cooperate with the research process
6. History of allergies or allergies to materials related to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic foot infection patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01-31 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of gene chips:Sensitivity, Specificity, Positive Predictive Value (PPV), NegativePredictive Value (NPV) | through study completion, an average of 1 year
The time (in minutes) taken for diagnosis using the gene chip method compared to the traditional method. | through study completion, an average of 1 year

SECONDARY OUTCOMES:
The time (in days) required for ulcer healing using the gene chip method compared to the traditional method. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- National Clinical Medical Research Center for Metabolic Diseases (Shanghai), Shanghai, China